CLINICAL TRIAL: NCT01853488
Title: Impact of Spinal Cord Injury on Bone Strength in Paralysed Extremities.
Brief Title: Bone Strength After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2010-13
Record Dates: First submitted 2013-05-02; First posted 2013-05-15 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2015-11

CONDITIONS: Spinal Cord Injury
Keywords: Osteoporosis; BMD; SCI; DXA; pQCT
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spinal Cord Injury: Persons with spinal cord injury Osteodensitometry DXA pQCT
  Interventions: Radiation: DXA; Radiation: pQCT
- Reference: Reference population (able-bodied) Osteodensitometry DXA pQCT
  Interventions: Radiation: DXA; Radiation: pQCT

INTERVENTIONS:
Radiation: DXA — Osteodensitometry
Radiation: pQCT — Osteodensitometry

SUMMARY:
Background:

After a traumatic spinal cord injury, a severe bone loss in the paralyzed extremities is observed. This leads to a osteoporosis which is connected to a high fracture risk.

Aims:

To compare the two measurement methods DEXA and pQCT concerning optimal diagnostics and assessment of fracture risk in subjects with spinal cord injury.

Subjects:

250 women and 250 men (age≥18, any AIS-classification) with an acute or chronic spinal cord injury will be recruited for this study. For a reference group, 500 able-bodied persons will be measured analogously.

Methods:

Using DEXA-Osteodensitometry, bone parameters of the lumbar vertebral column, proximal femur, distal radius, distal tibia and knee area will be assessed. Additionally, geometric bone parameters of the tibia will be measured by using pQCT. All measurements will be done unilaterally. For the assessment of potential risk factors for reduced bone stiffness after spinal cord injury a questionnaire will be used.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury
* mobilized patients
* written informed consent

Exclusion Criteria:

* current fracture
* limited mobility
* contractures of the lower limbs
* decubitus ulcer
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Swiss Paraplegic Centre Nottwil (in-patient or out-patient).
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2010-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Bone parameters | just one timepoint
  Measurement of the extremities with DEXA and pQCT

SECONDARY OUTCOMES:
Fractures | just one timepoint (questionnaire)
  Number of fractures since SCI

CONTACTS AND LOCATIONS:
Overall Officials: Angela Frotzler, PhD, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic-Centre, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- See also: Swiss Paraplegic Centre Nottwil — http://www.paranet.ch/en/pub/pan.htm